CLINICAL TRIAL: NCT01383096
Title: A Phase I Study To Investigate The Relative Bioavailability of OZ439 Formulations In Healthy Volunteers
Brief Title: Study To Investigate The Relative Bioavailability of OZ439 Formulations In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Nucleus Network Ltd (Other); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MMV_OZ439_11_001
Record Dates: First submitted 2011-06-23; First posted 2011-06-28 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Volunteers
Keywords: OZ439; Bioavailability; Food Effect
MeSH Terms: interventions — Powders; Suspensions; artefenomel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- Cohort 1 - Treatment A: OZ439 800mg PIB, fed (Active Comparator): OZ439 800 mg (as free base) as powder in a bottle (PIB)for reconstitution in a suspension prior to administration. Administered 30 minutes after a standard fatty breakfast.
  Interventions: Drug: OZ439 mesylate 800mg Powder in Bottle for Oral Suspension
- Cohort 1 - Treatment D: OZ439 800 mg Prototype F1 fasted (Experimental): OZ439 800 mg (as free base) as a prototype solution formulation 1. Administered fasted.
  Interventions: Drug: OZ439 mesylate 800mg Prototype Solution Formula 1
- Cohort 2 - Treatement H: OZ439 800 mg Prototype F2 fasted (Experimental): OZ439 800 mg (as free base) as a prototype solution formulation 2. Administered fasted.
  Interventions: Drug: OZ439 mesylate 800mg Prototype Solution Formula 2
- Cohort 3 - Treatement K: OZ439 400mg Prototype F1 fasted (Experimental): Best Prototype Solution - OZ439 400 mg as prototype solution formulation 1. Administered fasted.
  Interventions: Drug: OZ439 mesylate 400mg Prototype Solution Formula 1
- Cohort 1 - Treatement B: OZ439 800mg PIB fasted (Experimental): OZ439 800 mg (as free base) as powder in a bottle (PIB) for reconstitution in a suspension prior to oral administration. Administered fasted.
  Interventions: Drug: OZ439 mesylate 800mg Powder in Bottle for Oral Suspension
- Cohort 1 - Treatment C:OZ439 800mg PIB with milk (Experimental): OZ439 800 mg (as free base) as powder in a bottle (PIB) for reconstitution in a suspension prior to oral administration. Administered following 200 mL milk.
  Interventions: Drug: OZ439 mesylate 800mg Powder in Bottle for Oral Suspension
- Cohort 3 - Treatment J: OZ439 800mg Prototype F1 fasted (Experimental): Best Prototype Solution - OZ439 800 mg (as free base) as prototype solution formulation 1. Administered fasted.
  Interventions: Drug: OZ439 mesylate 800mg Prototype Solution Formula 1
- Cohort 1 - Treatement E: OZ439 800mg Prototype F1 with milk (Experimental): OZ439 800 mg (as free base) as a prototype solution formulation 1. Administered with milk.
  Interventions: Drug: OZ439 mesylate 800mg Prototype Solution Formula 1
- Cohort 2 - Treatement F: OZ439 800 mg PIB fasted (Experimental): OZ439 800 mg (as free base) as powder in a bottle (PIB) for reconstitution in a suspension prior to oral administration. Administered fasted.
  Interventions: Drug: OZ439 mesylate 800mg Powder in Bottle for Oral Suspension
- Cohort 2 - Treatement G: OZ439 800mg PIB with milk (Experimental): OZ439 800 mg (as free base) as powder in a bottle (PIB) for reconstitution in a suspension prior to oral administration. Administered following 200 mL milk.
  Interventions: Drug: OZ439 mesylate 800mg Powder in Bottle for Oral Suspension
- Cohort 2 - Treatement I: OZ349 800mg Prototype F2 with milk (Experimental): OZ439 800 mg (as free base) as a prototype solution formulation 2. Administered with milk.
  Interventions: Drug: OZ439 mesylate 800mg Prototype Solution Formula 2

INTERVENTIONS:
Drug: OZ439 mesylate 800mg Powder in Bottle for Oral Suspension — OZ439 800 mg (as free base) as powder in a bottle for reconstitution in a suspension prior to oral administration
  Other Names: OZ439 PIB
  Arms: Cohort 1 - Treatement B: OZ439 800mg PIB fasted; Cohort 1 - Treatment A: OZ439 800mg PIB, fed; Cohort 1 - Treatment C:OZ439 800mg PIB with milk; Cohort 2 - Treatement F: OZ439 800 mg PIB fasted; Cohort 2 - Treatement G: OZ439 800mg PIB with milk
Drug: OZ439 mesylate 400mg Prototype Solution Formula 1 — OZ439 400 mg (as free base) as a prototype solution formulation 1
  Other Names: OZ439 400mg Prototype 1
  Arms: Cohort 3 - Treatement K: OZ439 400mg Prototype F1 fasted
Drug: OZ439 mesylate 800mg Prototype Solution Formula 1 — OZ439 800 mg (as free base) as a prototype solution formulation 1
  Other Names: OZ439 800mg Prototype 1
  Arms: Cohort 1 - Treatement E: OZ439 800mg Prototype F1 with milk; Cohort 1 - Treatment D: OZ439 800 mg Prototype F1 fasted; Cohort 3 - Treatment J: OZ439 800mg Prototype F1 fasted
Drug: OZ439 mesylate 800mg Prototype Solution Formula 2 — OZ439 800 mg (as free base) as a prototype solution formulation 2
  Other Names: OZ439 800mg Prototype 2
  Arms: Cohort 2 - Treatement H: OZ439 800 mg Prototype F2 fasted; Cohort 2 - Treatement I: OZ349 800mg Prototype F2 with milk

SUMMARY:
This study is designed to assess prototype formulations compared to the aqueous dispersion of Active Pharmaceutical Ingredient used in Phase I and Phase IIa studies to date. It is hoped that the bioavailability of OZ439 can be enhanced in the fasted state to be close to that observed when given after food. This will improve the utility of OZ439 in the field as well as decreasing the cost of treatment (by decreasing the dose of OZ439 required) which is very important for an antimalarial drug product destined for use in developing counties.

DETAILED DESCRIPTION:
This study was a single centre, open-label, pharmacokinetic, randomized cross-over study in healthy male volunteers and post-menopausal women. This study was conducted over three different cohorts as follows:

Cohort 1: Subjects received a single 800 mg (as free base) dose of five different treatment regimes (treatments A, B, C, D and E) on five occasions.

Cohort 2: Subjects received a single 800 mg (as free base) dose of four different treatment regimes (treatments F, G, H and I) on four occasions.

Cohort 3: Subjects received a single dose, 800mg (as free base) of prototype solution formulation 1 (treatment J) and 400mg (as free base) of prototype solution formulation 1 (treatment K) on two occasions. The treatments were administered under the fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers between 18 and 55 years (inclusive). Post-menopausal women with amenorrhoea for at least 2 years are eligible confirmed by FSH level >/ = 25microlU/ml
* Body mass Index between 18 and 30 kg/m2, inclusive; and body weight > 50 kg.
* Healthy as determined by pre-study medical history, physical examination (including body temperature), 12 Lead ECG.
* Male volunteers must agree to use a double barrier method of contraception including abstinence, condom plus diaphragm or condom plus IUD or condom plus stable oral/transdermal/injectable hormonal contraceptive by female partner for at least 14 days prior to the time of the first dose of study drug through 90 days after the last dose of study drug and must also agree to not donate sperm for 90 days after the last dose of study drug. Vasectomy with zero sperm count for 6 months minimum prior to the first dose of study drug is an acceptable form of contraception
* Clinical laboratory tests at screening within the reference ranges or if outside the normal range not clinically significant. ALT, AST and total bilirubin must be within the normal range
* Able and willing to give written informed consent
* Willing and able to adhere to the lifestyle guideline requirements
* Willing and able to be confined to the Clinical Research Unit as required by the protocol

Exclusion Criteria:

* Evidence of or history of clinically significant oncologic, pulmonary, hepatic, cardiovascular, hematologic, metabolic, neurological, immunologic, nephrologic, endocrine, psychiatric disease, or current infection
* Evidence of or history of clinically significant gastrointestinal (excluding appendectomy and cholecystectomy) disease or current infection.
* Any condition that could possibly affect drug absorption, e.g. gastrectomy, diarrhea
* History of post-antibiotic colitis
* Pregnancy or breastfeeding
* QTc greater than 450 msec for males and females as corrected by the Fredricia's formula or evidence or history of abnormal cardiac rhythm
* History of drug or alcohol abuse within the past 2 years prior to Screening
* Tobacco users (includes stopping smoking less than 90 days prior to screening. "Tobacco use" includes smoking and the use of snuff and chewing tobacco, and other nicotine containing products
* Received an investigational drug or participated in another research study within 30 days of the first dose of study drug in any part of the study
* Use of prescription drugs within 14 days prior to the first dose of study drug in Period 1, or need for any antibiotic during the study
* Received any non prescription medications, vitamins, herbal supplements or dietary supplements within 7 days of the first dose of study drug in Period 1, unless prior approval is granted. Excluded from this list is intermittent use of acetaminophen at doses of up to 2 g/day
* Consumed alcohol within 72 hours of Day -1 in any part of the study, or have a positive alcohol screen at screening or each admission
* Consumed fruit juice or ate grapefruit within 7 days prior to the first dose of study drug in any part of the study
* Positive test for human immunodeficiency virus, hepatitis B surface antigen or anti-hepatitis C virus
* Positive urine drug screen at Screening or admission
* History of intolerance or hypersensitivity to artemisinins
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol
* Volunteers who have donated blood or experienced significant blood loss within 90 days of screening
* Hemoglobin < 13.5 g/dL for males and < 12.5 g/dL for females
* Any concern by the investigator regarding the safe participation of the volunteer or any reason the investigator considers the volunteer inappropriate for participation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Peter Hodsman, MD, Principal Investigator — AMREP Centre for Clinical Studies, Nucleus Network, 89 Commercial Road, Melbourne, VIC 3004 Australia
Locations (1):
- AMREP Centre for Clinical Studies, Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was randomised on 19-Apr-12; The last subject last visit was on 04-Aug-12. Subjects were recruited at the study site, Nucleus Network.
Pre-assignment Details: There was no wash-out, run-in or transition period between enrolment and group assignment.
Groups:
- Cohort 1: Subjects received a single dose of OZ439 800mg PIB Fed, then OZ439 PIB Fasted, then OZ439 800mg with milk, OZ439 800mg Prototype 1 Fasted, OZ439 800mg Prototype 1 with milk.
- Cohort 2: Subjects received a single of OZ439 800mg PIB Fasted, then OZ439 800mg with milk, OZ439 800mg Prototype 2 Fasted, OZ439 800mg Prototype 2 with milk.
- Cohort 3: Subjects received a 800mg single dose of OZ439 prototype solution formulation 1 fasted and then a 400mg single dose of OZ439 of prototype solution formulation 1 fasted.
Period: First Intervention (8 Days)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 19 | 17 | 16
Completed | 19 | 17 | 16
Not Completed | 0 | 0 | 0
Period: Second Intervention (8 Days)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 19 | 17 | 16
Completed | 19 | 16 | 14
Not Completed | 0 | 1 | 2
Not completed — Vomited Study Drug within 30min of admin | 0 | 0 | 1
Not completed — Haemoglobin was <13.5 g/dL | 0 | 1 | 1
Period: Third Intervention (8 Days)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 19 | 16 | 0 (Only 2 interventions in Cohort 3.)
Completed | 15 | 12 | 0 (Only 2 interventions in Cohort 3.)
Not Completed | 4 | 4 | 0
Not completed — Elevated AST | 0 | 1 | 0
Not completed — Vomited Study Drug within 30min of admin | 1 | 3 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — QTcF was greater than 450 msec | 1 | 0 | 0
Period: Fourth Intervention (8 Days)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 15 | 12 | 0 (Only 2 interventions in Cohort 3.)
Completed | 13 | 12 | 0 (Only 2 interventions in Cohort 3.)
Not Completed | 2 | 0 | 0
Not completed — Haemoglobin was <13.5 g/dL | 1 | 0 | 0
Not completed — QTcF was greater than 450 msec | 1 | 0 | 0
Period: Fifth Intervention (8 Days)
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 13 | 0 (Only 4 interventions in Cohort 2.) | 0 (Only 2 interventions in Cohort 3.)
Completed | 11 | 0 (Only 4 interventions in Cohort 2.) | 0 (Only 2 interventions in Cohort 3.)
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — haemoglobin was <13.5 g/dL | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population was comprised of all randomized subjects who received any amount of study drug and was based on the actual treatment received at each time point, if this differed from that to which the subject was randomized.
Groups:
- Cohort 2: Subjects received a single dose of OZ439 800mg PIB Fasted, then OZ439 800mg with milk, OZ439 800mg Prototype 2 Fasted, OZ439 800mg Prototype 2 with milk.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 19 | 17 | 16 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (6.2) | 27.2 (5.7) | 25.4 (4.4) | 27.4 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 19 | 17 | 16 | 52

OUTCOME MEASURES:

1. Primary Outcome: OZ439 Cmax
Description: The maximum observed plasma drug concentrations (Cmax)
Time Frame: 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 168 hours post dosing
Population: Pharmacokinetic Population: all subjects who received study drug, and completed at least one treatment (provided they had adequate OZ439 plasma concentration data) were included in the pharmacokinetic analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Cohort 1 - Treatment A: OZ439 800mg PIB Fed: OZ439 800 mg (as free base) as powder in a bottle (PIB) for reconstitution in a suspension prior to administration. Administered 30 minutes after a standard fatty breakfast.
- Cohort 1 - Treatment B: OZ439 800mg PIB Fasted; Cohort 2 - Treatment F: OZ439 800 mg PIB Fasted: OZ439 800 mg (as free base) as powder in a bottle (PIB) for reconstitution in a suspension prior to oral administration. Administered fasted.
- Cohort 1 - Treatment:OZ439 800mg PIB With Milk; Cohort 2 - Treatment G: OZ439 800mg PIB With Milk: OZ439 800 mg (as free base) as powder in a bottle (PIB) for reconstitution in a suspension prior to oral administration. Administered following 200 mL milk.
- Cohort 1 - Treatment E: OZ439 800mg Prototype F1 With Milk: OZ439 800 mg (as free base) as a prototype solution formulation 1. Administered with milk.
- Cohort 2 - Treatment H: OZ439 800 mg Prototype F2 Fasted: OZ439 800 mg (as free base) as a prototype solution formulation 2. Administered fasted.
- Cohort 2 - Treatment I: OZ349 800mg Prototype F2 With Milk: OZ439 800 mg (as free base) as a prototype solution formulation 2. Administered with milk.
- Cohort 3 - Treatment J: OZ439 800mg Prototype F1 Fasted: OZ439 800 mg (as free base) as prototype solution formulation 1. Administered fasted.
- Cohort 3 - Treatment K: OZ439 400mg Prototype F1 Fasted: OZ439 400 mg as prototype solution formulation 1. Administered fasted.
Arm/Group | Cohort 1 - Treatment A: OZ439 800mg PIB Fed | Cohort 1 - Treatment B: OZ439 800mg PIB Fasted | Cohort 1 - Treatment:OZ439 800mg PIB With Milk | Cohort 1 - Treatment D: OZ439 800 mg Prototype F1 Fasted | Cohort 1 - Treatment E: OZ439 800mg Prototype F1 With Milk | Cohort 2 - Treatment F: OZ439 800 mg PIB Fasted | Cohort 2 - Treatment G: OZ439 800mg PIB With Milk | Cohort 2 - Treatment H: OZ439 800 mg Prototype F2 Fasted | Cohort 2 - Treatment I: OZ349 800mg Prototype F2 With Milk | Cohort 3 - Treatment J: OZ439 800mg Prototype F1 Fasted | Cohort 3 - Treatment K: OZ439 400mg Prototype F1 Fasted
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 14 | 14
ng/ml | 1910 (32.9) | 827 (47.7) | 1930 (27.4) | 1440 (46.2) | 1830 (25.9) | 538 (33.2) | 1530 (31.2) | 846 (44.9) | 1680 (36.2) | 1160 (35.8) | 719 (29.0)

2. Primary Outcome: OZ439 AUC0-∞
Description: Area under the plasma concentration-time curve from zero to infinity (AUC0-∞)
Time Frame: 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 168 hours post dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng.h/mL
Groups:
- Cohort 1 - Treatement A: OZ439 800mg PIB Fed: OZ439 800 mg (as free base) as powder in a bottle (PIB) for reconstitution in a suspension prior to administration. Administered 30 minutes after a standard fatty breakfast.
- Cohort 1 - Treatement D: OZ439 800 mg Prototype F1 Fasted: OZ439 800 mg (as free base) as a prototype solution formulation 1. Administered fasted.
- Cohort 1 - Treatement E: OZ439 800mg Prototype F1 With Milk; Cohort 2 - Treatement I: OZ349 800mg Prototype F2 With Milk: OZ439 800 mg (as free base) as a prototype solution formulation 2. Administered with milk.
- Cohort 3 - Treatement J: OZ439 800mg Prototype F1 Fasted: OZ439 800 mg (as free base) as prototype solution formulation 1. Administered fasted.
- Cohort 3 - Treatement K: OZ439 400mg Prototype F1 Fasted: OZ439 400 mg as prototype solution formulation 1. Administered fasted.
Arm/Group | Cohort 1 - Treatement A: OZ439 800mg PIB Fed | Cohort 1 - Treatement B: OZ439 800mg PIB Fasted | Cohort 1 - Treatment C:OZ439 800mg PIB With Milk | Cohort 1 - Treatement D: OZ439 800 mg Prototype F1 Fasted | Cohort 1 - Treatement E: OZ439 800mg Prototype F1 With Milk | Cohort 2 - Treatement F: OZ439 800 mg PIB Fasted | Cohort 2 - Treatement G: OZ439 800mg PIB With Milk | Cohort 2 - Treatement H: OZ439 800 mg Prototype F2 Fasted | Cohort 2 - Treatement I: OZ349 800mg Prototype F2 With Milk | Cohort 3 - Treatement J: OZ439 800mg Prototype F1 Fasted | Cohort 3 - Treatement K: OZ439 400mg Prototype F1 Fasted
Number analyzed (Participants) | 11 | 12 | 11 | 11 | 11 | 10 | 12 | 12 | 12 | 14 | 14
ng.h/mL | 29200 (31.2) | 10700 (52.8) | 24500 (44.0) | 19000 (39.6) | 25800 (26.9) | 7460 (34.1) | 21600 (33.0) | 11700 (54.9) | 22900 (41.9) | 13800 (38.0) | 7410 (33.3)

3. Primary Outcome: OZ439 t1/2
Description: Apparent terminal half life (t1/2)
Time Frame: 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 168 hours post dosing
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Groups:
- Cohort 1 - Treatment C: OZ439 800mg PIB With Milk; Cohort 2 - Treatment G: OZ439 800mg PIB With Milk: OZ439 800 mg (as free base) as powder in a bottle (PIB) for reconstitution in a suspension prior to oral administration. Administered following 200 mL milk.
Arm/Group | Cohort 1 - Treatment A: OZ439 800mg PIB Fed | Cohort 1 - Treatment B: OZ439 800mg PIB Fasted | Cohort 1 - Treatment C: OZ439 800mg PIB With Milk | Cohort 1 - Treatment D: OZ439 800 mg Prototype F1 Fasted | Cohort 1 - Treatment E: OZ439 800mg Prototype F1 With Milk | Cohort 2 - Treatment F: OZ439 800 mg PIB Fasted | Cohort 2 - Treatment G: OZ439 800mg PIB With Milk | Cohort 2 - Treatment H: OZ439 800 mg Prototype F2 Fasted | Cohort 2 - Treatment I: OZ349 800mg Prototype F2 With Milk | Cohort 3 - Treatment J: OZ439 800mg Prototype F1 Fasted | Cohort 3 - Treatment K: OZ439 400mg Prototype F1 Fasted
Number analyzed (Participants) | 11 | 12 | 11 | 11 | 11 | 10 | 12 | 12 | 12 | 14 | 14
hours | 83.5 (27.8) | 82.3 (46.9) | 70.5 (45.9) | 90.0 (26.0) | 79.8 (27.2) | 84.7 (27.3) | 79.3 (28.0) | 85.7 (22.0) | 70.6 (17.7) | 63.6 (14.7) | 91.1 (35.7)

ADVERSE EVENTS:
Time Frame: Adverse event monitoring throughout the admission period.
Description: The Safety population was comprised of all randomised subjects who received any amount of study drug.
Arm/Group | Cohort 1 - Treatment A: OZ439 800mg PIB Fed | Cohort 1 - Treatment B: OZ439 800mg PIB Fasted | Cohort 1 - Treatment C: OZ439 800mg PIB With Milk | Cohort 1 - Treatment D: OZ439 800 mg Prototype F1 Fasted | Cohort 1 - Treatment E: OZ439 800mg Prototype F1 With Milk | Cohort 2 - Treatment F: OZ439 800 mg PIB Fasted | Cohort 2 - Treatment G: OZ439 800mg PIB With Milk | Cohort 2 - Treatment H: OZ439 800 mg Prototype F2 Fasted | Cohort 2 - Treatment I: OZ349 800mg Prototype F2 With Milk | Cohort 3 - Treatment J: OZ439 800mg Prototype F1 Fasted | Cohort 3 - Treatment K: OZ439 400mg Prototype F1 Fasted
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/14 | 0/15 | 0/17 | 0/15 | 0/13 | 0/15 | 0/17 | 0/13 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 5/17 | 5/14 | 4/15 | 8/17 | 9/15 | 5/13 | 4/15 | 12/17 | 5/13 | 10/14 | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - Treatment A: OZ439 800mg PIB Fed (N=17) | Cohort 1 - Treatment B: OZ439 800mg PIB Fasted (N=14) | Cohort 1 - Treatment C: OZ439 800mg PIB With Milk (N=15) | Cohort 1 - Treatment D: OZ439 800 mg Prototype F1 Fasted (N=17) | Cohort 1 - Treatment E: OZ439 800mg Prototype F1 With Milk (N=15) | Cohort 2 - Treatment F: OZ439 800 mg PIB Fasted (N=13) | Cohort 2 - Treatment G: OZ439 800mg PIB With Milk (N=15) | Cohort 2 - Treatment H: OZ439 800 mg Prototype F2 Fasted (N=17) | Cohort 2 - Treatment I: OZ349 800mg Prototype F2 With Milk (N=13) | Cohort 3 - Treatment J: OZ439 800mg Prototype F1 Fasted (N=14) | Cohort 3 - Treatment K: OZ439 400mg Prototype F1 Fasted (N=16)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 7 (7) | 5 (5) | 2 (2) | 2 (2) | 5 (5) | 4 (4) | 5 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (4) | 4 (4) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure orthostatic decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less